CLINICAL TRIAL: NCT06087913
Title: A Phase I Randomized, Placebo-controlled, Double-blind Study to Assess Safety, Pharmacokinetics, and Modeled Pharmacodynamics of a Vaginal Insert Containing Tenofovir Alafenamide and Elvitegravir
Brief Title: Safety and PK Multi-dose Study of TAF/EVG Vaginal Insert
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eastern Virginia Medical School (Other)
Collaborators: CONRAD (Other); University of Pittsburgh (Other); Centre for the AIDS Programme of Research in South Africa (Network); Kenya Medical Research Institute (Other); United States Agency for International Development (USAID) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MATRIX-001
Record Dates: First submitted 2023-09-07; First posted 2023-10-18 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Safety Issues
Keywords: vaginal insert; HIV; pre-exposure prophylaxis (PrEP)

STUDY DESIGN:
Intervention Model Description: Randomized, Placebo-Controlled, Double-Blind
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active (Experimental): TAF/EVG (20/16mg) vaginal insert
  Interventions: Drug: TAF/EVG vaginal insert
- Placebo (Placebo Comparator): Matching placebo insert
  Interventions: Drug: Matching Placebo vaginal insert

INTERVENTIONS:
Drug: TAF/EVG vaginal insert — vaginal insert applied daily for 3 days then every other day for 14 days
  Arms: Active
Drug: Matching Placebo vaginal insert — vaginal insert applied daily for 3 days then every other day for 14 days
  Arms: Placebo

SUMMARY:
MATRIX-001 will examine the safety, PK, modeled PD, and acceptability of inserts containing the combination of TAF and EVG applied vaginally, daily for 3 days, then every other day for 14 days. The inserts are ultimately intended to be the basis of an event-driven, on-demand method for prevention of HIV and HSV sexual infection.

DETAILED DESCRIPTION:
Participants will be enrolled across three sites, in USA, Kenya, and South Africa, approximately 20 per site. Participants will be randomized (1:1) to receive either a placebo or TAF/EVG vaginal insert as well as be randomized (1:1:1) to 3 different tissue sampling time points post-treatment (24hr, 48hr and 72hr after the last dose). Participants will be asked to complete 8 study visits with clinical and behavioral evaluations, and a subset will complete an in-depth interview to assess acceptability of vaginal insert use.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 50 years (inclusive) at Screening.
2. Assigned female sex at birth.
3. Able and willing to provide written informed consent to be screened for and enrolled in MATRIX-001 in one of the study languages (as specified in site SOP).
4. General good health (by volunteer history) without any evidence of clinically significant systemic disease (as determined by Investigator of Record [IoR] or designee).
5. Has had vaginal sex and has an intact uterus and cervix.
6. Has a regular and/or predictable bleeding pattern based on the opinion of the investigator, or is oligomenorrheic or amenorrhoeic.
7. HIV-uninfected based on testing performed at Screening and Enrollment (per protocol algorithms in Appendix II).
8. Negative urine pregnancy test at Screening and Enrollment.
9. Protected from pregnancy by an effective contraceptive method as confirmed by site SOP; effective methods include:

   * minimum of 3 months of use of a combined hormonal contraceptive method (except vaginal rings)
   * minimum of 6 months of use of a progestin only contraceptive method or copper IUD
   * Sterilization of participant or partner
   * Correct and consistent condom use (for US site only)
   * Abstinence from penile-vaginal intercourse (for US site only)
10. Participants over the age of 21 (inclusive) must have documentation of a Grade 0 Pap smear within the past 3 years prior to Enrollment, per the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 (Dated November 2007) to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017, or Grade 1 Pap smear at Screening with no treatment required.
11. Normal cervicovaginal mucosa (as defined in MATRIX-001 Study Specific Procedures [SSP] manual).
12. Willing and able to comply with protocol requirements, including abstaining from vaginal activity and product use at specified times.
13. Per participant report, if in a relationship, must be in a mutually monogamous relationship with a partner who is not known to be HIV positive or to currently have an STI.

Exclusion Criteria:

1. Per participant report, intends to do any of the following during the study participation period:

   * Become pregnant.
   * Breastfeed.
   * Relocate away from the study site.
   * Travel away from the study site for a time period that would interfere with product resupply and/or study participation.
2. Currently breastfeeding.
3. Positive HIV test at Screening or Enrollment.
4. History of sensitivity/allergy to any component of the study product, topical anesthetic, cellulose based thrombogenic material, or to both silver nitrate and Monsel's solution.
5. Positive test for Trichomonas vaginalis (TV), Neisseria gonorrhea (GC), Chlamydia trachomatis (CT), Treponema pallidum (Syphilis), or Hepatitis B surface antigen (HBsAg) at Screening or (per participant report) treated for GC, CT, TV, HBsAg or syphilis in the past 12 months.
6. Chronic or acute vulvar, vaginal or cervical symptoms (pain, irritation, spotting/bleeding other than what would be expected from contraceptive use, discharge, etc.).
7. Known bleeding/clotting disorder, including use of anti-coagulation.
8. Need for continued use of any contraindicated concomitant medications (as listed in Appendix III).
9. Participation in any other trial with use of an investigational drug/device within the last 30 days or planned participation in any other investigational trial with use of a drug/device during the study.
10. Participants who previously received an HIV vaccine or HIV broadly neutralizing antibody (bNAb) are not eligible. Individuals may be eligible if they participated in an HIV vaccine or bNAb study but have documentation that they did not receive active product (e.g., placebo recipients).
11. Prior use of PEP or oral PrEP (including FTC/TDF) in the past 4 weeks or any prior use of long-acting systemic PrEP (including cabotegravir or islatravir).
12. Grade 2 or higher pelvic finding or laboratory abnormality, per the DAIDS Table for Grading Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 and/or Addenda 1 (Female Genital Grading Tables for Use in Microbicide Studies [Dated November 2007]) or clinically significant laboratory abnormality as determined by the clinician.
13. Use of any of the following in the past 12 months: stimulants (cocaine [including crack], methamphetamine, or non-physician prescribed pharmaceutical-grade stimulants), or inhaled nitrates, or illicit injection drug use of any kind.
14. Has any other condition that, based on the opinion of the IoR or designee, would preclude provision of informed consent, make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-12-02 (Actual); Study Completion 2024-12-02 (Actual)

PRIMARY OUTCOMES:
Number and Severity of Adverse Events | Randomization through study completion, an average of 3 months
  Safety measured by reported AE's Grade 2 and higher

SECONDARY OUTCOMES:
Pharmacokinetics (PK) in cervicovaginal fluid (CVF) | through completion of study, an average of 3 months
  Concentrations of TFV, TAF and EVG
Pharmacokinetics (PK) in plasma | through completion of study, an average of 3 months
  Concentrations of TFV, TAF and EVG
Pharmacokinetics (PK) in cervicovaginal tissue | through completion of study, an average of 3 months
  Concentrations of TFV, TAF and EVG
Modeled in vitro Pharmacodynamics (PD) for HIV | Enrollment through study completion, an average of 3 months
  Rate of anti-viral activity in CVF
Modeled in vitro Pharmacodynamics (PD) for Herpes simplex virus (HSV) | Enrollment through study completion, an average of 3 months
  Rate of anti-viral activity in CVF
Number of participants who find using the vaginal insert acceptable. | Enrollment through study completion, an average of 3 months
  Responses to key questions on satisfaction, comfort with insertion, willingness to use the vaginal insert
Number of participants with changes to vaginal microbiome | Enrollment through study completion, an average of 3 months
  Evaluate mucosal factors and microbiome changes from baseline associated with mucosal function, including immune cells, pH, soluble markers, and immune cells.

OTHER OUTCOMES:
Modeled Tissue PD | Enrollment through study completion, an average of 3 months
  p24 antigen production in cervicovaginal tissue infected with HIV-1 ex vivo

CONTACTS AND LOCATIONS:
Overall Officials: Leila Mansoor, BPharm, PhD, Study Chair — Centre for the AIDS Programme of Research in South Africa; Nelly Mugo, MBChB, Study Chair — Kenya Medical Research Institute
Locations (3):
- Eastern Virginia Medical School Clinical Research Clinic (EVMS CRC), Norfolk, Virginia, United States
- Kenya Medical Research Institute (KEMRI), Thika, Kenya
- CAPRISA eThekwini Clinical Research Site, Durban, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dobard CW, Peet MM, Nishiura K, Holder A, Dinh C, Mitchell J, Khalil G, Pan Y, Singh ON, McCormick TJ, Agrahari V, Gupta P, Jonnalagadda S, Heneine W, Clark MR, Garcia-Lerma JG, Doncel GF. Single dose topical inserts containing tenofovir alafenamide fumarate and elvitegravir provide pre- and post-exposure protection against vaginal SHIV infection in macaques. EBioMedicine. 2022 Dec;86:104361. doi: 10.1016/j.ebiom.2022.104361. Epub 2022 Nov 21. PMID 36423375
- [Background] Thurman AR, Ouattara LA, Yousefieh N, Anderson PL, Bushman LR, Fang X, Hanif H, Clark M, Singh O, Doncel GF. A phase I study to assess safety, pharmacokinetics, and pharmacodynamics of a vaginal insert containing tenofovir alafenamide and elvitegravir. Front Cell Infect Microbiol. 2023 Apr 19;13:1130101. doi: 10.3389/fcimb.2023.1130101. eCollection 2023. PMID 37153145
- See also: MTN-039 Safety and PK of TAF/EVG rectal insert — https://clinicaltrials.gov/study/NCT04047420